CLINICAL TRIAL: NCT01759082
Title: The Angioma's Treatment Evaluation With Laser Doppler Imaging (LDI)
Acronym: TALDI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Tessa Mermod, Principal Investigator, University of Lausanne Hospitals
Other Study IDs: CHP
Record Dates: First submitted 2012-12-02; First posted 2013-01-02 (Estimated); Last update posted 2013-01-02 (Estimated); Status verified 2012-12

CONDITIONS: Port-wine Stains (PWS)
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Based on the Doppler effect, Laser Doppler Imaging (LDI) uses the interaction of light with moving erythrocytes to visualize perfusion in the microcirculatory system.

The new device to be used in this study have been adapted specifically for the application, facilitating its use in clinic. It has been designed to take a standard white light image of the area under inspection simultaneously with the perfusion image to facilitate clinical assessment.

Port-wine stain (PWS) birthmarks are congenital, low-flow vascular malformations of the skin found in approximately 0.3% of children. They are commonly found on the face and neck and may cause serious psychological consequences.

Lasers are the modality of choice for the treatment of PWS birthmarks. The use of PDL is very effective in PWS in closing the blood vessels and diminishing therefore the redness of the skin. Repeated laser treatment is necessary to achieve the desired clinical outcome.

Actually, the efficacy of the treatment of PWS by the laser is obtained by clinical inspection and digital photography.

By measuring the activity and intensity of the microcirculation present in and under the skin, the Laser-Doppler (LDI) will be capable of measuring the effect of Pulsed dye laser (PDL) treatment for port-wine stains.

ELIGIBILITY:
Inclusion Criteria:

* children aged 12 months to 6 years old
* port-wine stains (PWS)
* phototype's skin I, II or III

Exclusion Criteria:

* phototype's skin IV, V or VI
* prior treatment with laser
* contraindication of general anesthesia
* refusal from the parents

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Subjects presenting at the CHUV with PWS will be screened and their parents asked to join the study by a member of the research team.
  * Subjects who meet the inclusion criteria will be approached for informed written consent and enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Vascularization's percentage of the PWS with Laser Doppler | For each treatment, spaced about 2 months
  After the general anesthesia, we will take a measure before the treatment with the Laser Doppler of the vascularization's percentage of the PWS relative as the safe contralateral side.
  An other measure will be made after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DeBuys Roessingh, Dr MD PhD, Principal Investigator — Paediatrics Surgery